CLINICAL TRIAL: NCT05655988
Title: EVALUATION OF MESH MIGRATION THAT DO NOT REQUIRE FIXATION IN TOTAL EXTRAPERITONEAL INGUINAL HERNI REPAIR
Brief Title: MESH MIGRATION IN TOTAL EXTRAPERITONEAL INGUINAL HERNI REPAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Uzman Doktor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANILLERGİNNN
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; total extraperitoneal hernia repair; mesh migration; laparoscopic inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: After a total extraperitoneal inguinal hernia operation performed using a fixation-free mesh, ultrasonography will be performed on all patients to calculate the slip size of the mesh.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, the paramedic providing post-operative care, and the radiologist measuring the mesh migration will not know whether mesh fixation has been applied to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesh migration after TEPP / fixation free mesh (Active Comparator): After a total extraperitoneal inguinal hernia operation performed using a fixation-free mesh, ultrasonography will be performed on all patients to calculate the slip size of the mesh.
  Interventions: Diagnostic Test: inguinal ultrasonography
- mesh migration after TEPP / mesh with fixation (Active Comparator): TEPP surgeries performed with mesh fixation
  Interventions: Diagnostic Test: inguinal ultrasonography

INTERVENTIONS:
Diagnostic Test: inguinal ultrasonography — After a total extraperitoneal inguinal hernia operation performed using a fixation-free mesh, ultrasonography will be performed on all patients to calculate the slip size of the mesh.

SUMMARY:
Inguinal henri repair is among the most common operations performed by general surgery. The use of laparoscopy in inguinal hernia repair is becoming more common day by day. Laparoscopic inguinal hernia repair is being applied with increasing frequency due to its advantages such as reducing postoperative pain, providing early return to work and increasing patient satisfaction. Due to the widespread use of laparoscopic inguinal hernia repair, the best fixation method for the patches has become an increasingly questionable subject. It is thought that fixation of the patch with staples or clips may reduce the slippage of the patch, thus reducing the risk of hernia recurrence. In addition, it has been stated that the use of these fixation materials will both increase the cost and cause acute and chronic pain after surgery. In some studies in the literature, it was determined that not detecting the patch in laparoscopic inguinal hernia repair did not increase the recurrence. There are some studies showing that failure to fix the patch causes patch slippage in unilateral laparoscopic inguinal hernia repair. In this study, it was planned to investigate the rate of displacement of the patches fixed with staples in patches that do not require fixation in laparoscopic inguinal hernia repair surgeries, compared to the ones that were not fixed, and whether they cause recurrence. At the same time, whether the staples used for patch fixation increase postoperative pain will be evaluated with VAS (visual analog scale) at the postoperative 1st day, 1st month and 6th month after the operation, compared to the group without stapler patch fixation.

DETAILED DESCRIPTION:
72 patients who underwent laparoscopic inguinal hernia repair (Total Extraperitoneal repair) for unilateral inguinal hernia in Fatih Sultan Mehmet Training and Research Hospital General Surgery Clinic will be included in the study. The number of samples was calculated by performing impact power analysis. Informed consent form and voluntary consent form will be obtained from all patients.

A fixation-free patch (Medtronic Dextile Anatomical mesh, USA) will be used in all patients and the patients will be divided into 2 groups containing 36 patients. 1 patch fixation stapler will be placed on the pubic protrusion in the first group (Covidien ProTack Fixation Device 5mm, USA), no fixation material will be used in the second group. Randomization will be provided by determining which patient will be included in which group on the website www.randomiser.org. In all patients, 2 metallic clips (Covidien Endo Clip II Auto suture, USA) will be placed on the superomedial and inferomedial patch borders on the placed mesh, and patch slippage will be evaluated by determining the locations of the clips by superficial ultrasonography at the end of the surgery, at the 1st and 6th months after the surgery. Superficial USG will be performed by the researchers and no expense will be charged to the SSI. Visual Analogue Scale pain assessment questionnaire will be applied to all patients in the postoperative period and the results will be recorded. Patients will be evaluated in terms of inguinal hernia type (direct, indirect), age, gender, hernia size, previous lower abdomen surgery, and additional diseases. The surgeon and the patient performing the ultrasonographic evaluation will not know in which cases the patch has been detected, so the study will be designed as double-blind.

Patients with contraindicated general anesthesia, previous lower abdominal surgery, coagulopathy, iguinoscrotal hernia, incarcerated or strangulated hernia, with a lateral-medial hernia greater than 3 cm and a drain placed will not be included in the study.

Surgical technique: After the infraumbilical 1 cm camera trocar is placed, 2 5 mm working trocars will be inserted through the line alba. After the CO2 insufflation, a 30° camera will be used and the surgery will be performed under 12 mmHg CO2 pressure. After opening the preperitoneal area with the help of blunt dissection, the hernia sac will be clearly revealed and released. All patients will be evaluated peroperatively for the presence of direct and indirect hernia, by clearly demonstrating the spermatic cord structures and normal anatomy. Then, a fixation-free patch (Medtronic Dextile Anatomical Mesh, USA) will be placed on the defect area and fixed on the pubis in one group and not fixed in the other group. It will be ensured that the patch overflows at least 3-4 cm from the defect area. Before the patch is placed in the preperitoneal area, 3 pieces of 10 mm Medium Endo Clips (Covidien Endo Clip II Auto suture, USA) will be placed on the superomedial, inferolateral and inferomedial border. Then, after bleeding control, the layers will be closed in accordance with their anatomy.

The distances between the 3 clips placed at the end of the operation will be measured vertically and horizontally by USG and recorded as x and y values. Ultrasonographic evaluations of the patient will be performed by a surgeon trained in inguinal region Ultrasound.

During the statistical analysis, Mann-Whitney U, Student's T test, Pearson's Chi Square test and Fisher's test will be used where appropriate. Statistically significant p value will be taken into account when it is greater than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 18 years. patients who have not had previous inguinal region surgery. Patients with a direct and/or indirect hernia smaller than 5 cm.

Exclusion Criteria:

Complicated hernias. Patients undergoing mesh fixation for any reason. Patients with hemorrhage greater than 200 cc during or after surgery. Patients with drains. Patients with complications such as bleeding, early recurrence, wound infection in the early postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
mesh migration | 1 year
  Deciding whether these meshes really require detection based on the extent of migration in non-detection meshes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Patient data can be shared upon request.